CLINICAL TRIAL: NCT04972734
Title: Cohort of Premature Newborns for Charaterization of the Digestive Microbiota in Ulcerative Necrotizing Enterocolitis in Premature Infants
Acronym: CortECS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: MEDIS Laboratory (Unknown); QUAPA (Unknown); ENTeRisk (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2021 PONS
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Necrotizing Enterocolitis; Premature Birth
Keywords: Necrotizing Enterocolitis; prematurity; volatolomic and microbiological signatures; mast cell activation; blood tryptase assay; fungal digestive colonization; fecal calprotectin
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEC (Experimental): premature newborns developing a NEC
  Interventions: Biological: premature newborns developing a NEC
- Healthy control (Active Comparator): premature newborns without NEC
  Interventions: Biological: premature newborns without NEC

INTERVENTIONS:
Biological: premature newborns developing a NEC — weekly Blood sample and daily Stools sample during 12 weeks + Blood and stool sample during NEC
  Arms: NEC
Biological: premature newborns without NEC — weekly Blood sample and daily Stools sample during 12 weeks
  Arms: Healthy control

SUMMARY:
Compare the bacterial digestive microbiota during the stay in neonatal intensive care between a group of premature newborns developing a NEC (necrotizing enterocolitis) and a group of newborns free from NEC.

DETAILED DESCRIPTION:
Monitoring of a cohort of premature newborns with constitution of a collection of biological samples.

follow-up of newborns from birth up to 37 weeks of amenorrhea. The medical care of children will not be affected by their participation in the research.

* Sampling of amniotic fluid at the time of rupture of the water bag
* Sampling of the blood contained in the umbilical cord after clamping and section of the cord
* Sampling of meconium during the first 24 hours of life in intensive care / neonatal / maternity ward
* Collection of a daily stool sample until the end of hospitalization and when a NEC occurs
* Sampling of gastric residues during an episode of NEC
* Taking a daily sample of the newborn's enteral food
* Sampling of 500 µL of additional blood weekly during the punctures made for the treatment
* Daily statement of constants
* Record of all complications related to prematurity (HIV, bronchodysplastic, sepsis)

  * Blood analysis: CBC, platelets and CRP (data analyzed as part of the treatment). Specific analyzes for research will assess: the level of tryptase, IL4 and TLR4. The samples will be stored and analyzed in the immunology laboratory of the CHU Clermont Ferrand (Pr B. Evrard)
  * Analysis of the meconium sample and each stool emitted during hospitalization, and during an episode of ECUN

ELIGIBILITY:
Inclusion Criteria:

* born prematurely < 37 weeks of amenorrhea at the maternity ward of the CHU
* affiliated with a social security regime
* the holders of parental authority are able to give an informed consent to participate in the research

Exclusion Criteria:

* fetal pathology
* newborns whose holders of parental authority are under guardianship or under the age of 18
* refusal of participation by holders of parental authority

Ages: 1 Minute to 2 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
comparison of volatolomics results of the gut microbiota | Immediatly after the intervention
  Characterization of the gut microbiota using a capture method by hybridization of the gene encoding 16S rRNA
comparison of microbiological results of the gut microbiota | Immediatly after the intervention
  Characterization of the gut microbiota using a capture method by hybridization of the gene encoding 16S rRNA

SECONDARY OUTCOMES:
Fungal microbiota | Immediatly after the intervention
  Comparison of the fungal microbiota on 10 NECS and 10 healthy babies
Tryptasemia | Day 1, Day 3, Immediatly after the intervention
  measurement of blood tryptasemia
environmental xenobiotics | Day 1
  measurement of titane and silicia levels in placental and meconium assays
Milk protein composition | daily for 12 weekd
  milk protein determination
Milk lipid composition | daily for 12 weekd
  milk lipid determination

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No